CLINICAL TRIAL: NCT02723708
Title: Increasing Motivation in Attention Deficit Hyperactivity Disorder (ADHD) Via Self-activation of Ventral Tegmental Area (VTA)
Brief Title: Ventral Tegmental Area (VTA) Self-Activation in Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00070749; 1R01MH106751 (Other: NIMH)
Record Dates: First submitted 2016-03-24; First posted 2016-03-30 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Self activation of VTA bold signal (Experimental): Participants meeting study inclusion will then be scheduled for 4 fMRI sessions to assess and manipulate the ability to self-stimulate VTA activation. Each session will contain the same tasks and instructions. The experimental imaging task sessions will be done 24-72 hours apart and will consist of two types of runs: Test Runs (one pre-test and post-test each) and three Training Runs. Participants will be instructed to achieve heightened state of motivation using personally relevant thoughts and imagery.
  Interventions: Other: Real-Time functional Magnetic Resonance Imaging Feedback (RTFF)

INTERVENTIONS:
Other: Real-Time functional Magnetic Resonance Imaging Feedback (RTFF) — During the Activate trials, the thermometer will display the weighted average of VTA BOLD activation, dynamically updated every second. This continuously updated thermometer is the primary feedback mechanism.

SUMMARY:
The purpose of this study is to see if a non-medication intervention can increase motivation in individuals with ADHD by observing brain activity using magnetic resonance imaging (MRI).

DETAILED DESCRIPTION:
The study involves a screening visit and 4 experimental task sessions.During the screening visit subjects will undergo psychiatric screening to determine if they meet criteria for a diagnosis of ADHD. Participants who meet criteria for a diagnosis of ADHD will also have the following tests done at screening: breath alcohol test, urine drug screen and urine cotinine (by product of tobacco) screening and intelligence quotient (IQ) assessment. Eligible participants will complete a battery of cognitive assessments.

Participants meeting study inclusion will then be scheduled for 4 fMRI sessions to assess and manipulate the ability to self-stimulate VTA activation. Each session will contain the same tasks and instructions. The experimental imaging task sessions will be done within a one month window and will consist of two types of runs: Test Runs (one pre-test and post-test each) and three Training Runs.

The purpose of the Pre-Test is to establish a baseline level of self-generated VTA activation prior to receiving RTFF.

The Post-Test is designed to assess whether participants are better able to self-induce VTA BOLD signal in the absence of feedback (after receiving RTFF).

Participants will begin and end each scanning session with a 2-minute resting state scan. Participants will rest and fixate at a cross hair.

The purpose of the first run is to acquire data in functional space to facilitate registration of the VTA probabilistic atlas (MNI space) to functional space.

The Pre-Test and Post-Test runs will be identical and will have two trial types: Activate and Count.

During the Activate trials participants will be instructed to try to increase activity (BOLD signal) within their VTA. Specifically, we will instruct participants to try to get themselves into a heightened state of motivation using personally relevant thoughts and imagery. Importantly, they will be encouraged to optimize strategies for themselves.

During the Count trials, participants will be instructed to count backwards. The purpose of these trials is to: standardize the baseline period and to provide a distractor task to prevent engagement in activation strategies. There will be 5 repetitions of both trial types, separated by a jittered inter-trial-interval (ITI; total duration 4 minutes, 5 seconds).

The purpose of the subsequent training runs (n=3/day on each of the 4 days) is to provide participants with RTFF to assist them in increasing their VTA BOLD signal.

The training runs will consist of three trial types: Activate, Count, and Rest. For both Activate and Count Trials, participants will be given the same instructions as during the test runs. During the Rest trials participants will be instructed to rest and not think of anything in particular. The Activate and Rest trials will include a thermometer display, as described below. Each trial type will be repeated 5 times per run, separated by a jittered ITI (total duration 6 minutes, 18 seconds).

Following the Post-Test each day, the Cognitive Battery assessments will be repeated with the subject out of the scanner.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* Male or Female
* Confirmed diagnosis, any subtype as determined by the clinician administered Conner's Adult ADHD Diagnostic Interview for DSM-IV (CAADID) and clinical interview using the Mini International Neuropsychiatric Interview (MINI)
* T-Score > 65 on one of the DSM-IV relevant scales (Inattentive Symptoms, Hyperactive-Impulsive Symptoms, Total Symptoms or ADHD Index) on both the Self-Report and Observer versions of the Conner's Adult ADHD Rating Scales (CAARS)
* Cognitive functioning eaqual or greater than 80 as assessed by the Kaufman Brief Intelligence test, Second Edition (KBIT-II)

Exclusion Criteria:

* History of chronic/significant medical condition
* Current or past 6 month use of prescription medications for ADHD or other psychiatric condition
* Meets criteria for any other Axis I Disorder (determined the Mini International Neuropsychiatric Interview (MINI) other than nicotine dependence that is significantly impairing and would contraindicate participation in the present study
* Meets criteria for any Axis II Disorder
* Current substance abuse or dependence or history within the last 12 months; expired breath alcohol level > 0.0; Positive urine drug screen for any of the following: cannabis, amphetamines, opioids, benzodiazepines, barbiturates, cocaine
* Inability to understand written and/or spoken English language
* Claustrophobia or other contraindications to MRI scanning
* If female, pregnancy as determined by urine pregnancy test on each day of MRI scanning
* Presence of any metal in the body (e.g., implant, non-removable piercing, IUD)
* Head injury resulting in loss of consciousness
* Worked with metal (e.g., welding) or had an injury to the eye involving metal
* Weigh more than 250 pounds

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-08; Primary Completion 2021-10-05 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
Percent signal change in VTA BOLD activation | experiment session 1, approximately 1 hour
  The investigators will examine the % signal change in VTA BOLD activation during "Activate" versus "Count" trials during the Pre-Test run on experimental session 1, prior to RTFF training.
Change in VTA BOLD signal following RTFF | Baseline and following real time fMRI feedback, up to 4 weeks
  Four imaging task sessions will be done within a one month window

SECONDARY OUTCOMES:
Change in goal-directed behavior, as measured by the Effort discounting task | Baseline and following each of the RTFF sessions, up to 2 weeks
  The amount of time before the participant terminates will assess their willingness to persist in goal-directed behavior. Four task sessions will be done 24-72 hours apart
Change in inhibitory control, as measured by the Conners' Continuous Performance Task (CPT) | Baseline and following each of the RTFF sessions, up to 2 weeks
  Four task sessions will be done 24-72 hours apart
Change in attention, as measured by reaction time (RT) variability on the CPT | Baseline and following each of the RTFF sessions, up to 2 weeks
  Four task sessions will be done 24-72 hours apart

CONTACTS AND LOCATIONS:
Overall Officials: R. Alison Adcock, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke ADHD Program, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No